CLINICAL TRIAL: NCT05874492
Title: Evaluation of the Medical Benefit of a Spa Therapy on the Evolutionary Genius of Late Sequelae Fibrosis After Postoperative Radiotherapy for Breast Cancer in Remission
Brief Title: Evaluation of the Medical Benefit of Spa Therapy on Fibrosis After Postoperative Radiotherapy for Breast Cancer
Acronym: FIBROTHERME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Collaborators: Floralis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-A00091-44
Record Dates: First submitted 2023-04-13; First posted 2023-05-25 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Fibrosis; Breast Cancer
Keywords: fibrosis; breast cancer; radiotherapy; spa treatment
MeSH Terms: conditions — Fibrosis; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 2 groups:
  * Immediate spa therapy: the patient carries out the spa therapy soon after the enrolment in the study
  * Late spa therapy: the patient carries out the spa therapy after the 6-month follow up visit
Who Masked: Investigator
Masking Description: Randomisation will be carried out by the coordinating centre by telephone. This methodology will maintain the investigator's blindness, the coordinating centre will ask the patient not to talk to the investigator about her treatment during follow-up visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate spa treatment (Active Comparator): The spa treatment must be carried out within a maximum of 6 weeks after the inclusion visit.
  Interventions: Other: Thermal cure with a primary dermatological indication
- Late spa treatment (Sham Comparator): The spa treatment must be carried out after the 6-month visit.
  Interventions: Other: Thermal cure with a primary dermatological indication

INTERVENTIONS:
Other: Thermal cure with a primary dermatological indication — The thermal treatment combines baths which have a sedative, muscle-relaxing effect and encourage joint mobilisation, sprays which have a decongestant effect and, above all, thread-like showers which are carried out by jets of thermal water under high pressure for several minutes plus educational workshops (relaxation, sophrology, hygiene...)

SUMMARY:
FIBROTHERME is a comparative, controlled, randomized, multicenter and simple blinded (investigator) trial.

The aim of this study is to evaluate the medical benefit in terms of quality of life on the dermatological sequelae of fibrosis 6 months after a dermatologically oriented spa therapy in patients with severe late reactions affecting the skin and/or soft tissues at least 6 months after the end of postoperative radiotherapy for breast cancer.

DETAILED DESCRIPTION:
Radiation-induced fibrosis is an equivalent of an "orphan disease", in which oncologists have only recently shown interest, despite its prevalence. No study on the medical service provided by crenotherapy has been published in late radiation-induced fibrosis, which shares a common pathophysiology and medico-psycho-social sequelae with the sequelae of burns.

Chronic progressive dermatoses are part of the 12 main therapeutic orientations of medical thermalism. In particular, burn scars are a very current indication. Crenotherapy allows the attenuation, or even the disappearance of: pruritus and dysesthesia, local inflammation, hypertrophy and sclerosis and favours the recovery of chronic superficial erosions. Fibrous scars, even old ones, respond favourably to thermal treatments. The thermal treatment combines baths which have a sedative, muscle-relaxing effect and which favour joint mobilisation, sprays which have a decongestant effect and above all thread-like showers which are carried out by jets of thermal water under high pressure for several minutes.

The primary endpoint is the self-assessment by the patient of the dermatological quality of life by the DLQI score at 6 months after the end of the treatment compared between the intervention group (immediate treatment) and the control group (delayed treatment after 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 18 years
* In situ or invasive breast cancer
* DLQI ≥ 6 (at least moderate effect on patient's life)
* General status WHO 0-1
* Post-operative radiotherapy completed at least 6 months ago (with no maximum post radiotherapy delay)
* Unilateral breast radiotherapy
* Skin or soft tissue toxicity (- modules: Skin and subcutaneous tissue disorders / Musculoskeletal disorders / Reproductive organs and breast disorders) CTCAE v4.0 grade ≥ 2
* No inflammatory or infectious flare at inclusion
* Female of childbearing potential: negative urine pregnancy test at inclusion
* Patient informed and signed consent
* Affiliation to a social security systeme or equivalent

Exclusion Criteria:

* Progressive phase of cancer
* Metastatic disease
* Patient undergoing specific treatment for breast cancer (except adjuvant hormone therapy and/or adjuvant herceptin)
* Bilateral breast/parietal radiotherapy
* Breast prosthesis wearer
* Obvious skin ulceration in the treated breast
* Contraindication to spa treatment (acute inflammatory disease, active infections, heart failure with NYHA stage > 1, chronic respiratory failure, labile hypertension, bullous disease)
* Chronic progressive dermatological disease
* Women who are pregnant or likely to become pregnant within 6 months or who are breastfeeding
* Persons deprived of liberty or under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the medical benefit in terms of quality of life on the dermatological sequelae of fibrosis after a dermatologically oriented spa treatment. | 6 months
  Self-assessment by the patient of the dermatological quality of life by the DLQI (Dermatology Life Quality Index) score at 6 months after the end of the treatment compared between the intervention group (immediate treatment) and the control group (delayed treatment after 6 months). The DLQI score is between 0 and 30 where a high score indicates a significant impairment of quality of life.

SECONDARY OUTCOMES:
Generic quality of life | 6 months
  Evaluation of the medical benefit on generic quality of life. Patient self-assessment of generic quality of life using the EQ5D-3L. EQ-5D-3L is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ5D has 6 items intended to measure general health. The index score is between -0.53 and 1 where a high value indicates a good quality of life. The perceived health status is between 0 and 100 where a high value indicates good health.
Breast Cancer quality of life | 6 months
  Evaluation of the medical benefit on quality of life in patients with breast cancer. Patient self-assessment of quality of life using the EORTC (European Organisation for Research and Treatment of Cancer) QLQ C30 Score (Quality of Life of Cancer Patients). The EORTC QLQ-C30 has 15 domains. There is no total score. For each domain, the score is between 0 and 100 where a high score for overall health and functional dimensions represents a good quality of life; and a high score for symptomatic dimensions represents a high level of symptoms.
Senological quality of life | 6 months
  Evaluation of the medical benefit on the quality of senological life. Patient self-assessment of breast quality of life using the specific QLQ-BR23 module (breast cancer-specific quality of life questionnaire). The QLQ-BR23 has 8 domains. There is no total score. For each domain, the rank is between 1 and 5 where a high score represents the death.
Sequelae self assessment | 6 months
  Evaluation of the medical benefit on the self-assessment of the impact of radio induced sequelae. Self-assessment by the patient with an evaluation of the severity of the radiation-induced sequelae via the Pro-CTCAE self-questionnaire (item 25: skin dryness, item 28: itching, item 36: skin reaction to radiation, item 37: skin darkening, item 48: general pain, item 53: fatigue, item 54: anxiety, item 56: sadness, item 72: breast swelling and tenderness).
Lesions radiological assessment | 6 months
  Hetero-evaluation of the clinical and imaging efficacy of treatment on post-radiation lesions with CTCAE scale (Common Terminology Criteria for Adverse Events). For each domain, the score is between 0 and 100 where a high score for the functional dimensions represents a good quality of life; and a high score for the symptomatic dimensions represents a high level of symptoms.
Thickness radiological assessment | 6 months
  Hetero-evaluation of the clinical and imaging efficacy of treatment on post-radiation lesions of thickness. Imaging assessment with blinded measurement by an independent radiologist of comparative thickness by ultrasound: Dermal radiotoxicity can indeed be defined as the difference in dermal thickness between the 2 breasts (lesion area and mirror area of the contralateral breast) Dermal thickness is defined as the distance between the input ultrasound signal and the signal at the dermal-hypodermal interface at 6 months.
Volumetric aspect radiological assessment | 6 months
  Hetero-evaluation of the clinical and imaging efficacy of treatment on post-radiation lesions with HBCS (Harvard-Breast-Cosmesis-Scale). Evaluation of the cutaneous and volumetric aspect by an evaluation carried out by the practitioner with the Harvard-breast-cosmesis-scale (HBCS) score at 6 months. The HBCS score is assessed by a 4-point Likert scale where a high value indicates a high severity, 1 represents excellent breast shape or texture, 2 means good, 3 average and 4 poor with a severely deformed breast.
Consumption of treatment | 6 months
  Comparison of the type of treatment between the 2 groups.
Consumption of medical consultation | 6 months
  Comparison of the number of hospitalisations, consultations, physiotherapy, specific cosmetic consultations between the 2 groups.
Adverse events | 6 months
  Comparison of the adverse events in the 2 groups. Description of adverse events between the 2 groups.
Long-term cure quality of life benefice | 12 months
  Evaluation of the stability of the long-term effect for the immediate cure group. Evaluation of the maintenance of benefits at 12 months (stability of the long term effect) on the primary outcome and secondary outcomes. Self-assessment by the patient of the dermatological quality of life by the DLQI (Dermatology Life Quality Index).
Treatment effect size | 12 months
  Evaluation of the effect size of the treatment for the delayed treatment group. Confirmation of the size of the effect of the treatment on the primary and main secondary endpoints between 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Vogin, Principal Investigator — Centre François Baclesse
Locations (10):
- France (9):
  - Clinique Tivoli-Ducos, Bordeaux
  - Institut de Cancérologie de Bourgogne, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Institut Rafael, Levallois-Perret
  - Centre Azuréen de Cancérologie, Mougins
  - Centre Eugène Marquis, Rennes
  - Centre Hospitalier Roanne, Roanne
  - CHU Saint Etienne, Saint-Etienne
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
- Centre François Baclesse, Esch-sur-Alzette, Luxembourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Binder-Foucard F, Bossard N, Delafosse P, Belot A, Woronoff AS, Remontet L; French network of cancer registries (Francim). Cancer incidence and mortality in France over the 1980-2012 period: solid tumors. Rev Epidemiol Sante Publique. 2014 Apr;62(2):95-108. doi: 10.1016/j.respe.2013.11.073. Epub 2014 Mar 7. PMID 24613140
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] Mohanti BK, Bansal M. Late sequelae of radiotherapy in adults. Support Care Cancer. 2005 Oct;13(10):775-80. doi: 10.1007/s00520-004-0697-z. Epub 2005 Jul 22. PMID 16041503
- [Background] Burnet NG, Johansen J, Turesson I, Nyman J, Peacock JH. Describing patients' normal tissue reactions: concerning the possibility of individualising radiotherapy dose prescriptions based on potential predictive assays of normal tissue radiosensitivity. Steering Committee of the BioMed2 European Union Concerted Action Programme on the Development of Predictive Tests of Normal Tissue Response to Radiation Therapy. Int J Cancer. 1998 Dec 18;79(6):606-13. doi: 10.1002/(sici)1097-0215(19981218)79:63.0.co;2-y. PMID 9842969
- [Background] Johansson S, Svensson H, Denekamp J. Timescale of evolution of late radiation injury after postoperative radiotherapy of breast cancer patients. Int J Radiat Oncol Biol Phys. 2000 Oct 1;48(3):745-50. doi: 10.1016/s0360-3016(00)00674-x. PMID 11020571
- [Background] Sarin R, Dinshaw KA, Shrivastava SK, Sharma V, Deore SM. Therapeutic factors influencing the cosmetic outcome and late complications in the conservative management of early breast cancer. Int J Radiat Oncol Biol Phys. 1993 Sep 30;27(2):285-92. doi: 10.1016/0360-3016(93)90239-r. PMID 8407402
- [Background] Safwat A, Bentzen SM, Turesson I, Hendry JH. Deterministic rather than stochastic factors explain most of the variation in the expression of skin telangiectasia after radiotherapy. Int J Radiat Oncol Biol Phys. 2002 Jan 1;52(1):198-204. doi: 10.1016/s0360-3016(01)02690-6. PMID 11777639
- [Background] Foray N, Verrelle P. [DNA repair and repair diseases: between molecular models and clinical reality]. Bull Cancer. 2011 Mar;98(3):257-75. doi: 10.1684/bdc.2011.1326. French. PMID 21454154
- [Background] Yarnold J, Brotons MC. Pathogenetic mechanisms in radiation fibrosis. Radiother Oncol. 2010 Oct;97(1):149-61. doi: 10.1016/j.radonc.2010.09.002. Epub 2010 Sep 29. PMID 20888056
- [Background] Ly CL, Khetpal S, Heller DR, Higgins SA, Killelea B, Alperovich M, Avraham T. Comparing complications in irradiated and non-irradiated free-flaps in patients with bilateral immediate breast reconstruction and unilateral post-mastectomy radiotherapy. Microsurgery. 2021 Oct;41(7):615-621. doi: 10.1002/micr.30747. Epub 2021 Apr 22. PMID 33886127
- [Background] Offersen BV, Alsner J, Nielsen HM, Jakobsen EH, Nielsen MH, Krause M, Stenbygaard L, Mjaaland I, Schreiber A, Kasti UM, Overgaard J; Danish Breast Cancer Group Radiation Therapy Committee. Hypofractionated Versus Standard Fractionated Radiotherapy in Patients With Early Breast Cancer or Ductal Carcinoma In Situ in a Randomized Phase III Trial: The DBCG HYPO Trial. J Clin Oncol. 2020 Nov 1;38(31):3615-3625. doi: 10.1200/JCO.20.01363. Epub 2020 Sep 10. PMID 32910709
- [Background] Delanian S, Lefaix JL. Current management for late normal tissue injury: radiation-induced fibrosis and necrosis. Semin Radiat Oncol. 2007 Apr;17(2):99-107. doi: 10.1016/j.semradonc.2006.11.006. PMID 17395040
- [Background] Jacobson G, Bhatia S, Smith BJ, Button AM, Bodeker K, Buatti J. Randomized trial of pentoxifylline and vitamin E vs standard follow-up after breast irradiation to prevent breast fibrosis, evaluated by tissue compliance meter. Int J Radiat Oncol Biol Phys. 2013 Mar 1;85(3):604-8. doi: 10.1016/j.ijrobp.2012.06.042. Epub 2012 Jul 28. PMID 22846413
- [Background] Wong RK, Bensadoun RJ, Boers-Doets CB, Bryce J, Chan A, Epstein JB, Eaby-Sandy B, Lacouture ME. Clinical practice guidelines for the prevention and treatment of acute and late radiation reactions from the MASCC Skin Toxicity Study Group. Support Care Cancer. 2013 Oct;21(10):2933-48. doi: 10.1007/s00520-013-1896-2. Epub 2013 Aug 14. PMID 23942595
- [Background] Carl UM, Feldmeier JJ, Schmitt G, Hartmann KA. Hyperbaric oxygen therapy for late sequelae in women receiving radiation after breast-conserving surgery. Int J Radiat Oncol Biol Phys. 2001 Mar 15;49(4):1029-31. doi: 10.1016/s0360-3016(00)01515-7. PMID 11240244
- [Background] Hardy P. [Crenotherapy applied to scarring due to burns]. Ann Chir Plast. 1968 Jun;13(2):151-6. No abstract available. French. PMID 5678765
- [Background] Kwiatkowski F, Mouret-Reynier MA, Duclos M, Leger-Enreille A, Bridon F, Hahn T, Van Praagh-Doreau I, Travade A, Gironde M, Bezy O, Lecadet J, Vasson MP, Jouvency S, Cardinaud S, Roques CF, Bignon YJ. Long term improved quality of life by a 2-week group physical and educational intervention shortly after breast cancer chemotherapy completion. Results of the 'Programme of Accompanying women after breast Cancer treatment completion in Thermal resorts' (PACThe) randomised clinical trial of 251 patients. Eur J Cancer. 2013 May;49(7):1530-8. doi: 10.1016/j.ejca.2012.12.021. Epub 2013 Jan 24. PMID 23352440
- See also: Rapport 2013 de l'Observatoire sociétal des cancers. 2014. — https://www.ligue-cancer.net/sites/default/files/rapport-2013-observatoire-societal-des-cancers.pdf